CLINICAL TRIAL: NCT03423381
Title: Validation of a New Antidiabetic Food Concept Based on Modulation of the Gut Microbiota
Brief Title: Dietary Fibre and Metabolic Benefits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Vinnova (Other Government); Öste Venture AB (Unknown)
Responsible Party: Principal Investigator, Anne Nilsson, Associate professor, PhD, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-03575
Record Dates: First submitted 2017-12-29; First posted 2018-02-06 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Glucose Tolerance
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Crossover randomised
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cereal product 1 (Experimental): Cereal based müsli no. 1, made from typical Swedish cereals. All experimental products have different types and amounts of dietary fibre (df). The test portion is consumed as a single evening meal prior to determinations of test variables in the morning.
  Interventions: Other: Cereal product 1
- Cereal product 2 (Experimental): Cereal based muesli no. 2 made from typical Swedish cereals. All experimental products have different types and amounts of df. The test portion is consumed as a single evening meal prior to determinations of test variables in the morning.
  Interventions: Other: Cereal product 2
- Cereal product 3 (Experimental): Cereal based muesli no.3 made from typical Swedish cereals. All experimental products have different types and amounts of df.The test portion is consumed as a single evening meal prior to determinations of test variables in the morning.
  Interventions: Other: Cereal product 3
- Cereal product 4 (Experimental): Cereal based muesli no. 4 made from typical Swedish cereals. All experimental products have different types and amounts of df. The test portion is consumed as a single evening meal prior to determinations of test variables in the morning.
  Interventions: Other: Cereal product 4
- Cereal product 5 (Experimental): Cereal based muesli no. 5 made from typical Swedish cereals. All experimental products have different types and amounts of df. The test portion is consumed as a single evening meal prior to determinations of test variables in the morning.
  Interventions: Other: Cereal product 5
- Control product (Placebo Comparator): A cereal based product with low concentrations of df. The control portion is consumed as a single evening meal prior to determinations of test variables in the morning.
  Interventions: Other: Control product

INTERVENTIONS:
Other: Cereal product 1 — Cereal products based on rye, barley, wheat, oat, and corn
  Arms: Cereal product 1
Other: Cereal product 2 — Cereal products based on rye, barley, wheat, oat, and corn
  Arms: Cereal product 2
Other: Cereal product 3 — Cereal products based on rye, barley, wheat, oat, and corn
  Arms: Cereal product 3
Other: Cereal product 4 — Cereal products based on rye, barley, wheat, oat, and corn
  Arms: Cereal product 4
Other: Cereal product 5 — Cereal products based on rye, barley, wheat, oat, and corn
  Arms: Cereal product 5
Other: Control product — A cereal based product with low concentrations of df
  Arms: Control product

SUMMARY:
The aim of the project is to study the connection between bacterial fermentation in the colon of prebiotic substrates and effects on systemic metabolism and appetite i healthy humans

DETAILED DESCRIPTION:
The purpose with this project is to study the association between bacterial fermentation in the colon of specific mixtures of cereal dietary fiber and effects on systemic metabolism and appetite regulation. For this purpose, short term studies are performed in healthy adult subjects. Different cereals, cereal blends and from cereal extracted dietary fiber will be studied, as well as effects of different processing of the cereals. Cardiometabolic test markers and colonic fermentation metabolites will be followed up to 14 h after intake of the test substrates, and gut microbiota composition will be determined prior to and after the interventions.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults
* BMI<30
* non smokers
* consuming a non-vegetarian diet that follows the Nordic guidances

Exclusion Criteria:

* fasting blood glucose >6.1 mmol/L
* known cardio-metabolic disease (e.g. diabetes, hypertension, metabolic syndrome), gastro-intestinal disorders such as IBS (irritable bowel syndrome) that can interfere with the study results, food allergies. Further no antibiotics or probiotics should have been consumed within 4 weeks prior to and during the study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Blood glucose regulation | 0-14 h after intake
  Postprandial blood glucose regulation (incremental area under the curve) acute after intake of the test products and at forthcoming meals within 14 h after consumption of test products.

SECONDARY OUTCOMES:
serum insulin | 0-14 h after intake
  Postprandial serum insulin concentrations (incremental area under the curve) acute after intake of the test products and at forthcoming meals within 14 h after consumption of test products.
gut microbiota composition | first stool delivered from14 h after intake
  effects on gut microbiota composition after intake of prebiotics
plasma GLP-1 (glucagon-like peptide-1 ), PYY (peptide tyrosine tyrosine), Ghrelin | 0-14 h after intake
  Gastro-intestinale hormones involved in appetite and metabolic regulation
plasma: CRP (C reactive protein ), IL (interleukin)-6, IL-18, IL-8, IL-1, IL-10, LBP (lipopolysaccharide-binding protein), (PAI-1plasminogen activator inhibitor) | 0-14 h after intake
  Inflammatory markers in blood
plasma GLP-2 | 0-14 h after intake
  gut hormone involved in gut mucosa integrity
plasma SCFA (short-chain fatty acid) | 0-14 h after intake
  colonic fermentation metabolites
blood lipids | 0-14 h after intake
  cholesterol and free fatty acids in plasma
plasma adiponectin | 0-14 h after intake
  hormone involved in metabolic regulation
plasma BDNF (Brain-derived neurotrophic factor) | 0-14 h after intake
  signal protein important for brain functions, but also involved in metabolic regulation
plasma neurotensin | 0-14 h after intake
  a neuro peptide peptides involved in appetite and metabolic regulation
plasma Nesfatin-1 | 0-14 h after intake
  a neuro peptide that participates in the regulation of hunger and fat storage.

OTHER OUTCOMES:
Subjective appetite sensations | 0-14 h after intake
  determined with VAS (visual analogue scale) scales (0-100 mm)
mood (valence and activity) | 0-14 h after intake
  determined with VAS scales (0-100 mm)
Energy intake | 4 h after intake of a test product or the control product
  ad libitum intake at a second meal after intake of test products
breath hydrogen concentrations | 0-14 h after intake
  indicator of gut fermentation

CONTACTS AND LOCATIONS:
Overall Officials: Anne Nilsson, PhD, Principal Investigator — Food Technology, engineering, and Nutrition, LTH, Lund University
Locations (1):
- Food Technology, engineering and Nutrition, LTH, Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nilsson AC, Ostman EM, Knudsen KE, Holst JJ, Bjorck IM. A cereal-based evening meal rich in indigestible carbohydrates increases plasma butyrate the next morning. J Nutr. 2010 Nov;140(11):1932-6. doi: 10.3945/jn.110.123604. Epub 2010 Sep 1. PMID 20810606
- [Background] Nilsson AC, Johansson-Boll EV, Bjorck IM. Increased gut hormones and insulin sensitivity index following a 3-d intervention with a barley kernel-based product: a randomised cross-over study in healthy middle-aged subjects. Br J Nutr. 2015 Sep 28;114(6):899-907. doi: 10.1017/S0007114515002524. Epub 2015 Aug 11. PMID 26259632
- [Background] Kovatcheva-Datchary P, Nilsson A, Akrami R, Lee YS, De Vadder F, Arora T, Hallen A, Martens E, Bjorck I, Backhed F. Dietary Fiber-Induced Improvement in Glucose Metabolism Is Associated with Increased Abundance of Prevotella. Cell Metab. 2015 Dec 1;22(6):971-82. doi: 10.1016/j.cmet.2015.10.001. Epub 2015 Nov 6. PMID 26552345
- [Background] Sandberg JC, Bjorck IM, Nilsson AC. Rye-Based Evening Meals Favorably Affected Glucose Regulation and Appetite Variables at the Following Breakfast; A Randomized Controlled Study in Healthy Subjects. PLoS One. 2016 Mar 18;11(3):e0151985. doi: 10.1371/journal.pone.0151985. eCollection 2016. PMID 26990559
- [Background] Sandberg JC, Bjorck IME, Nilsson AC. Effects of whole grain rye, with and without resistant starch type 2 supplementation, on glucose tolerance, gut hormones, inflammation and appetite regulation in an 11-14.5 hour perspective; a randomized controlled study in healthy subjects. Nutr J. 2017 Apr 21;16(1):25. doi: 10.1186/s12937-017-0246-5. PMID 28431559
- [Background] Nilsson AC, Ostman EM, Holst JJ, Bjorck IM. Including indigestible carbohydrates in the evening meal of healthy subjects improves glucose tolerance, lowers inflammatory markers, and increases satiety after a subsequent standardized breakfast. J Nutr. 2008 Apr;138(4):732-9. doi: 10.1093/jn/138.4.732. PMID 18356328